CLINICAL TRIAL: NCT00278044
Title: Clinical Study and Gene Mutation Analysis of Adrenoleukodystrophy in Taiwanese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Fu Jen Catholic University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 94028
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-01

CONDITIONS: Adrenoleukodystrophy
Keywords: Search as text words in Annotation & Scope Note
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Blood Specimen Collection; Medical Records

INTERVENTIONS:
Procedure: blood sampling and medical records

SUMMARY:
Study the clinical manifestations and gene mutation of Taiwanese ALD patients

ELIGIBILITY:
Inclusion Criteria:

* X-ALD patients and family

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Study Completion 2007-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jao Shwann Liang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan